CLINICAL TRIAL: NCT07262736
Title: Pharmacokinetics of Clozapine and Norclozapine and the Effect of Pantoprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Orwa Albitar, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MY20090488
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers - Male and Female
MeSH Terms: interventions — Clozapine; Pantoprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clozapine (Active Comparator): Single dose of 12.5 mg clozapine
  Interventions: Drug: clozapine
- Clozapine and pantoprazole (Active Comparator): Single dose of 12.5 mg clozapine after five daily doses of pantoprazole tablets 40 mg to be started four days prior to the clozapine administration
  Interventions: Drug: clozapine; Drug: pantoprazole

INTERVENTIONS:
Drug: clozapine — Single dose of 12.5 mg clozapine (half 25 mg tablet)
Drug: pantoprazole — Five daily doses of pantoprazole tablets 40 mg to be started four days prior to the clozapine administration
  Arms: Clozapine and pantoprazole

SUMMARY:
Clozapine is an effective treatment for patients with schizophrenia who do not respond to other therapies, but its blood concentration varies widely between individuals due to genetic and physiological differences. Proton pump inhibitors such as pantoprazole are often prescribed in this population to prevent stomach discomfort, yet their impact on clozapine exposure has not been fully characterized. This clinical study will investigate the pharmacokinetics of clozapine and its main metabolite norclozapine, the influence of individual characteristics on drug exposure, and the effect of pantoprazole coadministration. Healthy adult volunteers will participate in a randomized open label cross over design, receiving a single dose of clozapine alone and again after pantoprazole treatment. Outcomes include clozapine and norclozapine plasma concentration time profiles, pharmacokinetic parameters, and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 18 to 50 years
2. No history of chronic medical or psychiatric disease, as confirmed by baseline medical evaluation, medical history, and electrocardiogram (ECG)
3. No use of any medications for at least two weeks before study initiation

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Current smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From pre-dose to 8 hours after a single oral dose of clozapine
  Maximum plasma concentration of clozapine following a single oral dose
Area Under the Plasma Concentration-Time Curve (AUC) | From pre-dose to 8 hours after dosing
  AUC of clozapine plasma concentration from time zero to the last measurable concentration following a single oral dose

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve Extrapolated to Infinity (AUCinf) | From pre-dose to last measurable concentration
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Time to Peak Concentration (Tmax) | From pre-dose to 8 hours after dosing
  Time to reach maximum observed plasma concentration of clozapine

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Sejahtera (Kesihatan & Pergigian), Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Albitar O, Muda MR, Ghadzi SMS, Noor DAM, Ibrahim B, Teh CH, Akkaif MA, Aziz FA. Pharmacogenetics and pharmacometabolomics predictors of clozapine and norclozapine pharmacokinetic exposure in healthy volunteers. Eur J Clin Pharmacol. 2025 Oct;81(10):1429-1438. doi: 10.1007/s00228-025-03884-w. Epub 2025 Jul 22. PMID 40694104
- [Result] Albitar O, Harun SN, Sheikh Ghadzi SM. Semi-physiological Pharmacokinetic Model of Clozapine and Norclozapine in Healthy, Non-smoking Volunteers: The Impact of Race and Genetics. CNS Drugs. 2024 Jul;38(7):571-581. doi: 10.1007/s40263-024-01092-1. Epub 2024 Jun 5. PMID 38836990